CLINICAL TRIAL: NCT07062497
Title: Ultrasound-guided Rectus Abdominis Muscle Sheath Block in Outpatient Umbilical Hernioplasties: a Comparative Analysis of the Use of Clonidine as an Adjuvant - Prospective Randomized Clinical Trial
Brief Title: Clonidine in Ultrasound-guided Rectus Sheath Block for Outpatient Umbilical Hernioplasty
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Samuel Navarro Abreu, MD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 83635224.9.0000.5259; 111111111111 (Other: REBEC)
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-12

CONDITIONS: Hernia, Umbilical; Clonidine; Pain, Postoperative; Ambulatory Surgical Procedures; Regional Anesthesia Block
Keywords: Rectus Sheath Block; Ultrasound-Guided Regional Anesthesia; Umbilical Hernia Repair; Clonidine; Local Anesthetics; Postoperative Pain Management; Ambulatory Surgery; Quality of Recovery; Alpha-2 Adrenergic Agonists; Pain Measurement; Analgesic Adjuvants
MeSH Terms: conditions — Hernia, Umbilical; Pain, Postoperative | interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: This is a parallel-assignment, randomized, double-blind, controlled clinical trial involving two intervention arms. Eligible adult patients undergoing ambulatory umbilical hernia repair are allocated in a 1:1 ratio to receive either ultrasound-guided rectus sheath block (RSB) with local anesthetics alone (control group) or RSB with local anesthetics plus clonidine (intervention group). Randomization is performed using block randomization with variable block sizes to ensure balance between groups. Allocation is concealed through sealed opaque envelopes. Both participants and outcome assessors are blinded to group assignment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectus Sheath Block (Active Comparator): Participants in this arm will receive bilateral ultrasound-guided rectus sheath block (RSB) without the addition of clonidine.
  Interventions: Drug: Rectus Sheath Block
- Rectus sheath block with clonidine (Active Comparator): Participants in this arm will receive bilateral ultrasound-guided rectus sheath block (RSB) with clonidine
  Interventions: Drug: Rectus Sheath Block with Clonidine

INTERVENTIONS:
Drug: Rectus Sheath Block — Participants in this arm will receive bilateral ultrasound-guided rectus sheath block (RSB) with a solution containing 8 mL of lidocaine 2% + 8 mL of ropivacaine 1%, diluted in 0.9% saline to a total volume of 20 mL, each side, without the addition of clonidine.
  Other Names: RSB
  Arms: Rectus Sheath Block
Drug: Rectus Sheath Block with Clonidine — Participants in this arm will receive bilateral ultrasound-guided rectus sheath block (RSB) with a solution containing 8 mL of lidocaine 2% + 8 mL of ropivacaine 1% + clonidine 75 mcg, diluted in 0.9% saline to a total volume of 20 mL, each side, without the addition of clonidine.
  Other Names: RSB with clonidine
  Arms: Rectus sheath block with clonidine

SUMMARY:
This clinical trial aims to evaluate the effectiveness of an ultrasound-guided nerve block technique as the sole anesthetic method for patients undergoing outpatient umbilical hernia surgery. The procedure, called rectus sheath block (RSB), involves injecting local anesthetic near the abdominal muscles to reduce pain during and after surgery. The study will compare two groups of adult patients: one receiving the nerve block with a medication called clonidine added to the anesthetic solution, and the other receiving the same block without clonidine. Clonidine may help improve pain control and reduce the need for additional pain medications. By analyzing pain scores, recovery quality, and potential side effects, the study seeks to determine whether the use of clonidine in this context is safe, cost-effective, and beneficial for patient recovery. Participants will answer questionnaires about their pain and recovery during the first 48 hours after surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, controlled clinical trial designed to evaluate the effectiveness and safety of adding clonidine to a local anesthetic solution for ultrasound-guided rectus sheath block (RSB) in adult patients undergoing ambulatory umbilical hernioplasty. The study will be conducted at the Ambulatory Surgery Unit of the Policlínica Universitária Piquet Carneiro, part of the Universidade do Estado do Rio de Janeiro (UERJ), between January 2025 and April 2026.

Eligible patients (ASA I or II, aged 18-65) scheduled for elective outpatient umbilical hernia repair with a hernial defect ≤ 4 cm will be randomized into two groups. The intervention group (BRA-CLO) will receive bilateral RSB with a solution containing 8 mL of lidocaine 2%, 8 mL of ropivacaine 1%, and clonidine 75 mcg, diluted in 0.9% saline to a total volume of 20 mL, administered on each side. The control group (BRA) will receive an identical volume and concentration of local anesthetic without the addition of clonidine.

RSB will be performed under real-time ultrasound guidance (Butterfly iQ+ probe) using an in-plane technique with a Quincke 22G needle. Sedation with midazolam, fentanyl, and propofol will be administered as required. The block will be performed preoperatively under standard monitoring, including ECG, pulse oximetry, and non-invasive blood pressure.

The primary hypothesis is that the addition of clonidine will enhance the quality of intraoperative and postoperative analgesia, reduce opioid consumption, and improve overall postoperative recovery without increasing the risk of adverse events. To assess recovery quality, the validated Quality of Recovery-15 (QoR-15) questionnaire will be administered at postoperative 24 and 48 hours. Pain will be assessed using the Numeric Rating Scale (NRS) at predefined intervals (PACU, 24h and 48h). Sedation will be measured with the Richmond Agitation-Sedation Scale (RASS), and adverse events such as bradycardia, nausea, vomiting, conversion to general anesthesia, and postoperative complications will be recorded.

Randomization will be performed using block randomization with variable block sizes (4, 6, or 8) generated in R (v4.4.1), and allocation concealment will be ensured with sealed opaque envelopes. Data will be collected and managed using the REDCap platform, ensuring confidentiality and integrity.

The study aims to fill an important gap in evidence regarding the use of alpha-2 adrenergic agonists as adjuvants in abdominal wall blocks, especially in the context of ambulatory surgery. It is expected that the findings will support the safe and effective use of clonidine to optimize regional anesthesia protocols in hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years;
* Both male and female participants;
* ASA physical status I or II (American Society of Anesthesiologists classification);
* Scheduled for elective ambulatory umbilical hernia repair;
* Hernial defect size ≤ 4 cm (small to medium).

Exclusion Criteria:

* Refusal or inability to provide written informed consent;
* Cognitive or psychiatric disorders that impair comprehension or adherence to the study protocol;
* Known allergy or hypersensitivity to local anesthetics, clonidine, opioids, nonsteroidal anti-inflammatory drugs (NSAIDs), or other analgesics;
* Participation in another clinical trial within the previous 30 days;
* Missing data or loss to follow-up during postoperative assessments;
* Contraindications to regional anesthesia or known coagulopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Total opioid postoperative consumption | 48 hours postoperative
  Total amount of opioid analgesics (in milligrams of tramadol equivalents) administered from the end of the surgical procedure to 48 hours postoperatively.
Postoperative pain intensity assessed by Numeric Rating Scale (NRS) | At post-anesthesia care unit (PACU) admission (immediately after surgery), 24 hours after surgery, and 48 hours after surgery.
  Pain scores reported by the patient using the 11-point Numeric Rating Scale (0 = no pain; 10 = worst imaginable pain) at each time point.
Total intraoperative opioid consumption | From induction of anesthesia to the end of surgery.
  Total intraoperative fentanyl consumption

SECONDARY OUTCOMES:
Quality of recovery assessed by QoR-15 questionnaire | At post-anesthesia care unit (PACU) admission (immediately after surgery), 24 hours after surgery, and 48 hours after surgery.
  Patient-reported recovery quality measured using the Quality of Recovery-15 (QoR-15) instrument, scored from 0 to 150, with higher scores indicating better recovery.
Incidence of postoperative nausea and vomiting (PONV) | 48 hours postoperatively
  Number of patients who experience at least one episode of nausea and/or vomiting in the first 48 hours after surgery.

OTHER OUTCOMES:
Postoperative Richmond Agitation-Sedation Scale (RASS) sedation score | At post-anesthesia care unit (PACU) admission (immediately after surgery).
  The Richmond Agitation-Sedation Scale (RASS) is a 10-point scale used to assess the level of sedation and agitation in patients. The scale ranges from -5 (unarousable) to +4 (combative), where higher positive scores indicate higher levels of agitation (worse outcome), and lower negative scores indicate deeper sedation (also considered a worse outcome depending on clinical context). A score of 0 corresponds to an alert and calm patient, which is considered optimal.
Bradycardia | From the start of surgery until discharge from the post-anesthesia care unit (PACU), 2 hours after surgery.
  Incidence of bradycardia
Hypotension | From the start of surgery until discharge from the post-anesthesia care unit (PACU), 2 hours after surgery.
  Incidence of hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinica Universitária Piquet Carneiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon reasonable request to the corresponding author, following appropriate de-identification procedures and in accordance with local ethical guidelines.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Individual participant data (IPD) and supporting information will be made available beginning 6 months after publication of the primary results and will remain available for 5 years after publication.
Access Criteria: Access to the de-identified individual participant data and supporting documents will be granted to qualified researchers upon reasonable request, provided that the proposed use is for scientific research purposes and complies with institutional and ethical guidelines. Requests should be submitted to the corresponding author and will be evaluated by the research team. Data will be shared under a data use agreement.

REFERENCES:
- [Background] Cucchiaro G, Ganesh A. The effects of clonidine on postoperative analgesia after peripheral nerve blockade in children. Anesth Analg. 2007 Mar;104(3):532-7. doi: 10.1213/01.ane.0000253548.97479.b8. PMID 17312203
- [Background] Xuan C, Yan W, Wang D, Li C, Ma H, Mueller A, Wang J. The Facilitatory Effects of Adjuvant Pharmaceutics to Prolong the Duration of Local Anesthetic for Peripheral Nerve Block: A Systematic Review and Network Meta-analysis. Anesth Analg. 2021 Sep 1;133(3):620-629. doi: 10.1213/ANE.0000000000005640. PMID 34153021
- [Background] Visoiu M, Scholz S, Malek MM, Carullo PC. The addition of clonidine to ropivacaine in rectus sheath nerve blocks for pediatric patients undergoing laparoscopic appendectomy: A double blinded randomized prospective study. J Clin Anesth. 2021 Aug;71:110254. doi: 10.1016/j.jclinane.2021.110254. Epub 2021 Mar 19. PMID 33752119
- [Background] Kwon HJ, Kim YJ, Kim Y, Kim S, Cho H, Lee JH, Kim DH, Jeong SM. Complications and Technical Consideration of Ultrasound-Guided Rectus Sheath Blocks: A Retrospective Analysis of 4033 Patients. Anesth Analg. 2023 Feb 1;136(2):365-372. doi: 10.1213/ANE.0000000000006282. Epub 2022 Nov 29. PMID 36638514